CLINICAL TRIAL: NCT02124707
Title: LCCC 1330 - A Phase II Study of Weekly Carboplatin, Paclitaxel and Cetuximab for Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Weekly Carboplatin, Paclitaxel and Cetuximab Treatment for Patients With Recurrent or Metastatic SCCHN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1330
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma of the Head and Neck
Keywords: Head and neck cancer; Squamous cell carcinoma; Metastatic; Recurrent; Phase II; Carboplatin; Paclitaxel; Cetuximab
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell; Neoplasm Metastasis; Recurrence | interventions — Cetuximab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin, Paclitaxel and Cetuximab (Experimental): A 6 week course of weekly carboplatin, paclitaxel, and cetuximab will be administered to 38 patients with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN). Once protocol therapy is complete, cetuximab may be continued if the patient and physician agree. Within 3 weeks of the end of protocol therapy, response will be assessed, and if the patient has achieved at least stable disease, the treating physician may continue to treat with weekly cetuximab at their discretion until disease progression. Patients will be followed for a maximum of 3 years after the end of the 6 week treatment phase.
  Interventions: Drug: Cetuximab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Cetuximab — 400mg/m2 IV (in the vein) on day 1 of week 1 and 250mg/m2 IV (in the vein) on day 1 of weeks 2-6. Patients with stable disease may continue on maintenance therapy at the 250mg/m2 dose until disease progression.
  Other Names: Erbitux
Drug: Paclitaxel — 135mg/m2 IV (in the vein) on day 1 of each 1 week for 6 weeks.
  Other Names: Taxol
Drug: Carboplatin — AUC2, IV (in the vein) on day 1 of each 1 week for 6 weeks.
  Other Names: Paraplatin

SUMMARY:
This is a non-randomized, open-label phase II trial of 38 patients with recurrent or metastatic SCCHN. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 with good organ function and will be treated with six weekly cycles of carboplatin, paclitaxel and cetuximab. Following assessment of response, the treating physician at their discretion may continue to treat with weekly cetuximab as maintenance until disease progression. The study is designed to evaluate whether this regimen improves median overall survival (OS) as compared to an historical control population treated with a platinum plus 5-fluorouracil (5-FU). There is currently no agreed upon first line therapy for recurrent or metastatic SCCHN; regimen options are highly toxic, inconvenient and resource intensive. Our study regimen has been used extensively for induction therapy and off-protocol in palliative care, but treatment outcomes have yet to be defined by a clinical trial.

DETAILED DESCRIPTION:
Because of their high response rates and low toxicity, the taxane, carboplatin, cetuximab regimens have frequently been adapted for use in the palliative setting. At UNC, we have observed high rates of response, leading to symptomatic benefit and low toxicity. Further, the regimen de-medicalizes the patient's life in several important ways. First, unlike with the EXTREME regimen, no PORT or 4 day infusion is required. Second, the regimen gives only six weeks of cytotoxic therapy. Finally, in our experience there is a low rate of severe toxicity and this, coupled with the high rate of response, may improve quality of life. We are not aware of any presented or published results on the use of this combination in palliative therapy; with the adoption of this regimen in clinical practice, documentation of its benefit via conduct of a clinical trial is needed.

We propose a study designed to detect an improvement in median OS versus a historical control. The control arm from the EXTREME trial achieved a median OS of 7.4 months. We hypothesize that a less toxic and more effective 3-drug regimen will result in improved median OS compared with the control arm from EXTREME (median 7.4 months). The toxicity associated with EXTREME is primarily attributable to the cisplatin and 5FU cytotoxic backbone as its toxicity has been consistent in multiple studies of both palliative therapy and induction therapy. If a 4-month improvement in OS is achieved with acceptable toxicity, we will consider this regimen worth of further study.

Secondary objectives will include characterizing changes in quality of life (QoL), symptoms and toxicities. Patients will be encouraged to co-enroll into the UNCseq protocol for further exploration of associations between genetic changes and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Histologically or cytologically confirmed recurrent or metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN). All primary sites are eligible excluding WHO type III or EBV nasopharyngeal (WHO type I and WHO type II allowed as long as they are EBV negative)
* ECOG performance status 0-1
* Adequate organ and marrow function as defined below. Laboratory tests should be completed within 14 days prior to registration: ANC greater than or equal to 1,500/mm3, Platelets greater than or equal to 100,000/mm3, HgB greater than 9g/dL (acceptable to reach this by transfusion), Total bilirubin less than or equal to 1.5mg/dL, Albumin greater than 2.5 g/dL, AST(SGOT)/ALT(SGPT) less than or equal to 2.5X institutional upper limit of normal, alkaline phosphatase less than or equal to 2.5 x upper limit of normal, GFR greater than 30 mL/min (by standard Cockroft and Gault formula or measured via 24 hour urine collection)
* Women of childbearing potential (WOCBP) with negative serum or urine pregnancy test within 7 days of D1 of treatment
* WOCBP and men must agree to use adequate contraception prior to study entry and for duration of treatment under this protocol; adequate contraception is defined as any medically recommended method (or combination of methods) per standard of care.
* Cancer must be considered incurable by the treating clinician
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* History of prior cumulative exposure to > 300mg/m2 cisplatin, AUC of 18 of carboplatin, or their combined equivalent within one year prior to enrollment
* Surgery or radiation within the four weeks prior to D1 of treatment under this protocol
* Prior systemic chemotherapy unless it was part of definitive-intent (curative intent) treatment more than 6 months before study entry
* Other active, invasive malignancy requiring ongoing therapy or expected to require systemic therapy within two years; localized squamous cell carcinoma of the skin, basal-cell carcinoma of the skin, carcinoma in-situ of the cervix, or other malignancies requiring locally ablative therapy only will not result in exclusion
* Pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Bon Secours Virginia Health System, Midlothian, Virginia

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://www.unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the University of North Carolina at Chapel Hill Hospitals and Bon Secours Virginia Health System June 16, 2014 to February 27, 2017
Pre-assignment Details: Nineteen subjects were consented to this trial. Of these, 3 were not eligible, 2 withdrew before treatment. 14 subjects were treated.
Groups:
- Carboplatin, Paclitaxel and Cetuximab: A 6 week course of weekly carboplatin, paclitaxel, and cetuximab will be administered to 38 patients with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN). Cetuximab may be continued if the patient and physician agree. Within 3 weeks of the end of protocol therapy, response will be assessed, and if the patient has achieved at least stable disease, the treating physician may continue to treat with weekly cetuximab at their discretion until disease progression. Patients will be followed for a maximum of 3 years after the end of the 6 week treatment phase.
  Cetuximab: 400mg/m2 IV (in the vein) on day 1 of week 1 and 250mg/m2 IV (in the vein) on day 1 of weeks 2-6. Patients with stable disease may continue at the 250mg/m2 dose until disease progression.
  Paclitaxel: 135mg/m2 IV (in the vein) on day 1 of each 1 week for 6 weeks.
  Carboplatin: Squared Area under the curve (AUC2), IV (in the vein) on day 1 of each 1 week for 6 week
Period: Overall Study
Arm/Group | Carboplatin, Paclitaxel and Cetuximab
Started | 14
Completed | 7
Not Completed | 7
Not completed — Adverse Event | 5
Not completed — Physician Decision | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Carboplatin, Paclitaxel and Cetuximab: A 6 week course of weekly carboplatin, paclitaxel, and cetuximab will be administered to 38 patients with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN). Cetuximab may be continued if the patient and physician agree. Within 3 weeks of the end of protocol therapy, response will be assessed, and if the patient has achieved at least stable disease, the treating physician may continue to treat with weekly cetuximab at their discretion until disease progression. Patients will be followed for a maximum of 3 years after the end of the 6 week treatment phase.
  Cetuximab: 400mg/m2 IV (in the vein) on day 1 of week 1 and 250mg/m2 IV (in the vein) on day 1 of weeks 2-6. Patients with stable disease may continue at the 250mg/m2 dose until disease progression.
  Paclitaxel: 135mg/m2 IV (in the vein) on day 1 of each 1 week for 6 weeks.
  Carboplatin: AUC2, IV (in the vein) on day 1 of each 1 week for 6 week
Arm/Group | Carboplatin, Paclitaxel and Cetuximab
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] — Age range of treated subjects
  years | 62 [26 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 14
Primary Tumor Site [Count of Participants; unit: Participants]
  Glottis | 1
  Hypopharynx | 1
  Lymph Nodes | 1
  Oral Cavity | 7
  Ororpharynx | 4
T Stage [Count of Participants; unit: Participants] — Per the American Joint Committee on Cancer(AJCC) Staging Manual 7th edition; T stage describes features of a primary tumor including size, depth of invasion, perineural invasion, tumor grade, anatomic location, and skull involvement where lower number = lower risk and X = not evaluable.
  Participants
    Tx | 2
    T1 | 1
    T2 | 5
    T3 | 2
    T4a | 4
N Stage [Count of Participants; unit: Participants] — A count of participants, staged per the American Joint Committee on Cancer (AJCC) Staging Manual 7th edition. N stage is a nodal assessment including size, number of involved lymph nodes, location of nodes where lower number = lower risk and x = not evaluable.
  Participants
    N0 | 3
    N1 | 1
    N2b | 8
    Nx | 1
    Not reported | 1
M Stage [Count of Participants; unit: Participants] — Metastasis staged per the American Joint Committee on Cancer (AJCC) Staging Manual 7th edition; M0 is no distant metastasis (lower risk) and M1 is distant metastasis present
  Participants
    M0 | 8
    M1 | 6
human papillomavirus (HPV) infection status [Count of Participants; unit: Participants] — positive results are better.
  Participants
    Negative | 4
    Positive | 5
    Unknown | 5
P16 [Count of Participants; unit: Participants] — P16 is a protein; positive results are better.
  Participants
    Negative | 5
    Positive | 5
    Unknown | 4

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival
Description: Overall survival after treatment with weekly carboplatin, paclitaxel and cetuximab for 6 weeks with or without the addition of maintenance weekly cetuximab is defined as the time from D1 of treatment under this protocol until death as a result of any cause.
Time Frame: 36 months
Population: Two patients who received treatment were not analyzed after they withdrew from the study.
Measure: Median (Full Range); unit: Days
Groups:
- Carboplatin, Paclitaxel and Cetuximab: A 6 week course of weekly carboplatin, paclitaxel, and cetuximab will be administered to 38 patients with recurrent or metastatic SCCHN. Once protocol therapy is complete, cetuximab may be continued if the patient and physician agree. Within 3 weeks of the end of protocol therapy, response will be assessed, and if the patient has achieved at least stable disease, the treating physician may continue to treat with weekly cetuximab at their discretion until disease progression. Patients will be followed for a maximum of 3 years after the end of the 6 week treatment phase.
  Cetuximab: 400mg/m2 IV (in the vein) on day 1 of week 1 and 250mg/m2 IV (in the vein) on day 1 of weeks 2-6. Patients with stable disease may continue on maintenance therapy at the 250mg/m2 dose until disease progression.
  Paclitaxel: 135mg/m2 IV (in the vein) on day 1 of each 1 week for 6 weeks.
  Carboplatin: AUC2, IV (in the vein) on day 1 of each 1 week for 6 week
Arm/Group | Carboplatin, Paclitaxel and Cetuximab
Number analyzed (Participants) | 12
Days | 231 [89 to 700]

2. Secondary Outcome: Median Progression Free Survival
Description: Progression events will be defined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions Progression free survival after treatment with weekly carboplatin, paclitaxel and cetuximab for 6 weeks with or without the addition of maintenance weekly cetuximab is defined as the time from Day 1 of treatment until progression or death as a result of any cause.
Time Frame: 36 months
Population: Two patients who received treatment were not analyzed after they withdrew from the study.
Measure: Median (Full Range); unit: Days
Groups:
- Carboplatin, Paclitaxel and Cetuximab: A 6 week course of weekly carboplatin, paclitaxel, and cetuximab will be administered to 38 patients with recurrent or metastatic SCCHN. Once protocol therapy is complete, cetuximab may be continued if the patient and physician agree. Within 3 weeks of the end of protocol therapy, response will be assessed, and if the patient has achieved at least stable disease, the treating physician may continue to treat with weekly cetuximab at their discretion until disease progression. Patients will be followed for a maximum of 3 years after the end of the 6 week treatment phase.
  Cetuximab: 400mg/m2 IV (in the vein) on day 1 of week 1 and 250mg/m2 IV (in the vein) on day 1 of weeks 2-6. Patients with stable disease may continue on maintenance therapy at the 250mg/m2 dose until disease progression.
  Paclitaxel: 135mg/m2 IV (in the vein) on day 1 of each 1 week for 6 weeks.
  Carboplatin: AUC2, IV (in the vein) on day 1 of each 1 week for 6 weeks.
Arm/Group | Carboplatin, Paclitaxel and Cetuximab
Number analyzed (Participants) | 12
Days | 132 [89 to 392]

3. Secondary Outcome: Overall Response Rate by Participants
Description: Number of complete response (CR) and partial response (PR) after study treatment with weekly carboplatin, paclitaxel, and cetuximab for 6 weeks. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT scan: CR is defined as disappearance of all target lesions; and PR as >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: 6 weeks
Population: Two patients who received treatment were not analyzed after they withdrew from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin, Paclitaxel and Cetuximab
Number analyzed (Participants) | 12
Participants
  CR | 1
  PR | 6
  Neither CR nor PR | 5

4. Secondary Outcome: Incidence of Adverse Events
Description: Grade 3 and 4 toxicities associated with this combined chemotherapy regimen as assessed by clinician assessment using the NCI Common Terminology Criteria for Adverse Events,a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care Activities of daily living (ADL). Grade 4 Life-threatening consequences; urgent intervention indicated. Describe patient reported symptoms associated with this regimen.
Time Frame: 18 weeks
Measure: Number; unit: incidents
Arm/Group | Carboplatin, Paclitaxel and Cetuximab
Number analyzed (Participants) | 14
incidents
  Small Intestinal Obstruction | 1
  Fatigue | 2
  Gait Disturbance | 1
  Infusion Related Reaction | 1
  Sepsis | 1
  Lymphocyte Count Decreased | 3
  Neutrophil Count Decreased | 6
  Platelet Count Decreased | 1
  White Blood Cell Decreased | 7
  Hypernatremia | 1
  Hypoalbuminemia | 1
  Hypomagnesemia | 1
  Myalgia | 1
  Pneumothorax | 1
  Dry Skin | 1
  Rash Acneiform | 5

5. Secondary Outcome: Head and Neck Quality of Life Assessments
Description: Quality of life (QOL) as measured by the Functional Assessment of Cancer Therapy - Head and Neck (FACT-HN) questionnaire. The FACT-HN is the FACT-General (FACT-G) and a head and neck cancer specific, 12 item subscale given at baseline, at end of treatment, and at first follow-up visit. The FACT-G is a 27 item measure of general QOL assessing function in 4 domains: physical well-being (PWB), social-family well-being (SFWB), emotional well-being (EWB) and functional well-being (FWB). Items are rated by patients on a Likert scale from 0 to 4, with all subscales summed to give a total score with a range of 0-148 Higher scores represent better QOL.
Time Frame: Baseline, End of treatment (EOT), First follow-up visit (8-12 weeks after EOT)
Population: Two patients who received treatment did not complete the measures at any timepoint.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Carboplatin, Paclitaxel and Cetuximab
Number analyzed (Participants) | 12
score on a scale
  QOL at Baseline | 92.5 [63 to 129]
  QOL at End of Treatment | 87 [64 to 113]
  QOL at First Follow-up | 88 [63 to 121]

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Carboplatin, Paclitaxel and Cetuximab
All-Cause Mortality (participants affected / at risk) | 12/14
Serious Adverse Events (participants affected / at risk) | 6/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin, Paclitaxel and Cetuximab (N=14)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Infusion related reaction (General disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin, Paclitaxel and Cetuximab (N=14)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Agitation (Psychiatric disorders) | 1
Alanine aminotransferase incre (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 11
Anorexia (Metabolism and nutrition disorders) | 2
Anxiety (Psychiatric disorders) | 1
Aspartate aminotransferase inc (Investigations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Catheter related infection (Infections and infestations) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 2
Confusion (Psychiatric disorders) | 1
Conjunctivitis (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine increased (Investigations) | 2
Diarrhea (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema limbs (General disorders) | 1
Enterocolitis infectious (Infections and infestations) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 3
Gait disturbance (General disorders) | 1
Gastrointestinal disorders - O (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 5
Infusion related reaction (General disorders) | 1
Insomnia (Psychiatric disorders) | 2
Libido decreased (Psychiatric disorders) | 1
Localized edema (General disorders) | 1
Lymphedema (Vascular disorders) | 2
Lymphocyte count decreased (Investigations) | 7
Mucositis oral (Gastrointestinal disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Neutrophil count decreased (Investigations) | 10
Obstruction gastric (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 5
Proctitis (Gastrointestinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 10
Sepsis (Infections and infestations) | 1
Sinus tachycardia (Cardiac disorders) | 1
Skin and subcutaneous tissue d (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Urinary frequency (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 2
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT02124707/Prot_SAP_000.pdf